CLINICAL TRIAL: NCT06998459
Title: Evaluation of the Effectiveness of Bian-Stone Therapy in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Shu-Yu Yang, Director of the Department of Pediatrics, Division of Traditional Chinese Medicine, Taichung Tzu Chi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC 111-13
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Evaluation of Bian Stone Therapy for Autism Spectrum Disorder
Keywords: Bian-Stone therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bian-Stone therapy (Experimental): Once a week, each session lasting 30 minutes, for a duration of six months.
  Interventions: Other: Bian-Stone therapy
- control group (Placebo Comparator): Maintain the original treatment approach
  Interventions: Other: Maintain the original treatment approach

INTERVENTIONS:
Other: Bian-Stone therapy — Once a week, each session lasting 30 minutes, for a duration of six months.
  Arms: Bian-Stone therapy
Other: Maintain the original treatment approach — Maintain the original treatment approach
  Arms: control group

SUMMARY:
Autism spectrum disorder (ASD) is a pervasive developmental disorder of brain abnormalities. It presents with difficulties of communication and social interaction, and restrictive interests and restrictive behaviors. The CDC suggested that the popularity of ASD people is 1.5% in the US, and the male to female ratio is 4.5 to 1. In Taiwan, the popularity is around 1%, with the number increasing in recent years.

The exact etiology of ASD has remained unknown. Currently, the treatments include behavioral therapies, medication and alternative therapies. However, there is no specific way to cure the core symptoms of ASD. This study plans to apply behavioral therapies and traditional Chinese medical Bian-stone therapies on ASD children and compare the results between ASD children with only behavioral therapies. We will record theAutism Behavior Checklist-Taiwan Version, Development Screening Chart for Children Aged 0-6 Years, and Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) before and after the treatments, and meanwhile using the Ryodoraku Measurement (良導絡) to measure the meridian energy. This study aims to evaluate the effectiveness of traditional Chinese medical Bian-stone therapies in ASD children. In addition, we hope to investigate the relationship between ASD symptoms and twelve meridians and assess the patterns in Chinese medicine. Hopefully this study will help strengthen the clinical evidence in TCM treatments for ASD children and improve the efficacy of this disease.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed with Autism Spectrum Disorder (ASD) based on DSM-5 diagnostic criteria, and additionally screened using the T-STAT assessment tool, with severity categorized as mild or moderate.

  2.Patients aged between 1.5 and under 6 years, regardless of gender. 3.A Full-Scale IQ of 70 or above as measured by the Wechsler Intelligence Scale for Children (WISC).

  4.No prior experience with Bianshi therapy. 5.Consent obtained from the patient or their guardian to provide relevant clinical data for use in this study.

Exclusion Criteria:

* 1.Individuals who do not meet the aforementioned inclusion criteria. 2.Severe hearing, visual, or motor impairments, or diagnoses of cerebral palsy or epilepsy.

  3.Presence of other comorbid conditions, such as Tuberous Sclerosis, Fragile X Syndrome, Timothy Syndrome, male Rett Syndrome (with MECP2 gene mutation), and other chromosomal abnormalities (e.g., Angelman syndrome, Prader-Willi syndrome, Phelan-McDermid syndrome, and other related syndromes).

  4.Use of dietary supplements or health products.

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Autism Behavior Checklist-Taiwan Version | Pre-test, mid-test at 3 months, and post-test at 6 months.
  This checklist includes 47 items across five categories: sensory, relating, body and object use, language, and social and self-help skills. The raw score is based on the number of questions answered "yes." This score is then compared with appropriate norms to determine the individual's position relative to the norms.
  Pre-test, mid-test at 3 months, and post-test at 6 months. Development Screening Chart for Children Aged 0-6 Years This scale measures development across five categories: communication and language development, social and personality development, gross motor skills, fine motor skills, and perceptual and cognitive development. It includes 19 age groups, from birth to 72 months, and organizes developmental abilities in order.
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) | Pre-test, mid-test at 3 months, and post-test at 6 months.
  This tool assesses adaptive behavior across four domains: communication, daily living skills, socialization, and motor skills. It provides standard scores for each domain and an overall composite score, with lower scores indicating higher levels of impairment. Age-equivalent scores for each domain were calculated by averaging the subdomain scores, based on previous research methodologies.
Development Screening Chart for Children Aged 0-6 Years | Pre-test, mid-test at 3 months, and post-test at 6 months.
  This scale measures development across five categories: communication and language development, social and personality development, gross motor skills, fine motor skills, and perceptual and cognitive development. It includes 19 age groups, from birth to 72 months, and organizes developmental abilities in order.

SECONDARY OUTCOMES:
Meridian Energy Analysis Device | Pre-test, mid-test at 3 months, and post-test at 6 months.
  This study used the MEAD Meridian Energy Analysis Device (ME-10), developed by Med-Pex, Taipei, Taiwan, and certified by the Department of Health (Medical Device No. 002062). Based on Dr. Yoshio Nakatani's Ryodoraku theory, the device measures Qi imbalances across 24 points on the 12 major meridians. Measured acupoints included LU9, PC7, HT7, SI4, SJ4, LI5, ST42, LR3, KI4, BL65, GB40, and SP3. Qi imbalance patterns in allergic rhinitis participants were analyzed by comparing mean meridian values. The upper/lower ratio, calculated by dividing the sum of upper meridian values by that of the lower, reflects mental health status.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Yang, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taichung Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes